CLINICAL TRIAL: NCT06620809
Title: An Open-Label Exploratory Clinical Trial to Assess the Safety and Efficacy of NouvSoma001 in the Treatment of Neuromyelitis Optica Spectrum Disorders
Brief Title: The Safety and Efficacy of NouvSoma001 in Neuromyelitis Optica Spectrum Disorders
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: iRegene Therapeutics Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Wei Wang, Prof., Tongji Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NouvSoma001inNMOSD
Record Dates: First submitted 2024-09-22; First posted 2024-10-01 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Neuromyelitis Optica Spectrum Disorders
Keywords: Neuromyelitis Optica Spectrum Disorders; extracelluar vesicles
MeSH Terms: conditions — Neuromyelitis Optica | interventions — Injections, Spinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extracellular vesicles group (Experimental): Patients in this group will receive extracellular vesicles derived from human-induced neural stem cells for intrathecal injection once a day for 1 day.
  Interventions: Drug: Extracellular vesicles derived from human-induced neural stem cells for intrathecal injection
- Extracellular vesicles placebo group (Placebo Comparator): Patients in this group will receive a placebo of extracellular vesicles derived from human-induced neural stem cells for intrathecal injection once a day for 1 day.
  Interventions: Drug: A placebo of extracellular vesicles derived from human-induced neural stem cells for intrathecal injection

INTERVENTIONS:
Drug: Extracellular vesicles derived from human-induced neural stem cells for intrathecal injection — Extracellular vesicles derived from human-induced neural stem cells for intrathecal injection（5×10^9 particles）
  Other Names: NouvSoma001
  Arms: Extracellular vesicles group
Drug: A placebo of extracellular vesicles derived from human-induced neural stem cells for intrathecal injection — Extracellular vesicles placebo(5×10^9 particles）
  Other Names: NouvSoma001
  Arms: Extracellular vesicles placebo group

SUMMARY:
This is a single-center, randomized, open-label, placebo-controlled, dose-escalation trial. The objective of this research is to evaluate the safety, tolerability, and efficacy of intrathecal administration of human-induced neural stem cell-derived extracellular vesicles (NouvSoma001) for the treatment of neuromyelitis optica spectrum disorders.

DETAILED DESCRIPTION:
This is a single-center, randomized, open-label, placebo-controlled, dose-escalation trial. The study consists of two parts: Part 1 is a dose-escalation study, while Part 2 is a dose-extension study based on the results of Part 1. Part 1 will follow a traditional 3+3 dose-escalation design, enrolling a total of 9 subjects. In Cohort 1, participants will receive 5 × 10^9 particles; in Cohort 2, they will receive 1.5 × 10^10 particles; and in Cohort 3, they will receive 3 × 10^10 particles. If no dose-limiting toxicities (DLTs) are observed within 2 weeks after the initial administration, a new cohort will be enrolled at the next higher dose level. If DLTs are observed in 1 participant, another 2 participants will be treated at the same dose level. Dose escalation will cease if DLTs are observed in more than 33% of the participants. In Part 2, the remaining 60 participants will be randomized in a 2:1 ratio to the treatment and placebo groups, with the dose level determined by the Data Safety Monitoring Board based on the results of Part 1.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must meet the 2015 International Consensus Diagnostic Criteria for Neuromyelitis Optica Spectrum Disorder (NMOSD) and test positive for AQP4 antibodies.
2. Symptom onset occurred within 7 days prior to enrollment, with associated severe pain, lower limb motor dysfunction, or urinary/bowel impairment.
3. Males or Females aged between 18 and 65 years.
4. The Expanded Disability Status Scale (EDSS) score prior to the current disease episode is ≤ 4.
5. Female participants of childbearing potential must present a negative pregnancy test at screening and agree to use effective contraception throughout the study period.
6. Informed consent must be obtained from the patient or their legal representative, with a signed consent form must be provided.

Exclusion Criteria:

1. Abnormal laboratory indicators of the subjects need to be excluded, including, but not limited to, the following indicators:

   White Blood Cell Count <3*10^9/L Neutrophil Count <1.5*10^9/L <1.5*10^9/L Hemoglobin <85 <85 g/L Platelet Count <80*10^9/L <80*10^9/L Serum Creatinine >1.5*ULN Total Bilirubin >1.5*ULN AST (GOT) >3*ULN ALT (GPT) >3*ULN Alkaline Phosphatase >2*ULN (AST = Aspartate Aminotransferase; GOT = Glutamic-Oxaloacetic Transaminase; ALT = Alanine Aminotransferase; GPT = Glutamic-Pyruvic Transaminase)
2. Any contraindications to lumbar puncture.
3. Pregnant or breastfeeding women, and patients with plans to conceive during the trial.
4. Patients with a known history of allergies to human-derived biological products or those with an allergic predisposition.
5. Patients who have undergone hematopoietic stem cell transplantation or lymphatic irradiation before enrollment.
6. Patients who have participated in any other clinical trial within the last 3 months.
7. Patients with severe comorbidities, including immunodeficiency or coagulation disorders.
8. Patients with active suicidal ideation within 6 months before screening or have a history of suicide attempts within 3 years before screening.
9. Patients with severe psychiatric symptoms that prevent clinical cooperation.
10. Patients with positive for alcohol addiction or drug abuse.
11. Patients with malignant tumors.
12. Patients who have experienced any of the following events within 12 weeks before enrollment: myocardial infarction, unstable ischemic heart disease, stroke, or New York Heart Association Class IV heart failure.
13. Patients with persistent systemic infections and severe local infections.
14. Patients unable to undergo magnetic resonance imaging during the trial.
15. Patients deemed unsuitable for participation by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of all adverse events (AE) and serious adverse events (SAE) | Up to 6 month after treatment initiation
  The assessment of adverse events and serious adverse events

SECONDARY OUTCOMES:
The incidence and severity of all adverse events (AE) and serious adverse events (SAE) | Up to 18 month after treatment initiation
  The assessment of adverse events and serious adverse events
Magnetic Resonance Imaging（MRI）scan of the brain and spinal cord at month 3、6 | Up to 6 month after treatment initiation
The score of Visual analogue scale（VAS） at month 1、3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
Brief Pain Inventory - Short form (BPI-SF) at month 1、3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
The score of Expanded Disability Status Scale （EDSS） at month 1、3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
  The score of EDSS ranges from 0 to 10, and 10 represents the worst.
The score of Fecal Incontinence Severity Index (FISI) at month 1、3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
  The score of FISI ranges from 0 to 3, and 3 represents the worst.
The score of Hauser Ambulance Index （contains The timed 25-foot walk）at month 1、3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
  The score of HAI ranges from 1 to 11, and 11 represents the worst.
The score of Hamilton Despression Scale at month 1、3、6 compared with baseline and control group | Up to 6 month after treatment initiation
  The score of Hamilton Depression Scale ranges from 0 to 81, and 81 represents the worst
The score of Hamilton Anxiety Scale at month 1、3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
  The score of Hamilton Anxiety Scale ranges from 0 to 56, and 56 represents the worst.
The Modified Rankin Scale (mRS) | Up to 6 month after treatment initiation
  To assess mRS of subjects within month 1、3、6 after treatment initiation
The value of Quality of Life (EQ-5D-5L) at month 1、3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
The incidence of Columbia-Suicide Severity Rating Scale (C-SSRS) events at month 1、3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
The value of Nfl、GFAP in the serum at month 1、3、6 compared with baseline and control group | Up to 6 month after treatment initiation
The value of white blood cell count in cerebrospinal fluid at month 3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
The value of QAlb in cerebrospinal fluid at month 3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
The value of Nfl in cerebrospinal fluid at month 3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
The value of GFAP in cerebrospinal fluid at month 3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
The value of IL-1β in cerebrospinal fluid at month 3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
The value of IL-6 in cerebrospinal fluid at month 3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
The value of TNF-α in cerebrospinal fluid at month 3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
The value of sTREM2 in cerebrospinal fluid at month 3、6 compared with baseline and control group. | Up to 6 month after treatment initiation
Examination of visual function at month 1、3、6 | Up to 6 month after treatment initiation
  Orbital MRI and VEP (Visual evoked potential)
Optical coherence tomography (OCT) at month 3、6 | Up to 6 month after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Dai-shi Tian, MD, Principal Investigator — Tongji Hospoital; Wei Wang, MD, Principal Investigator — Tongji Hospoital; Chuan Qin, MD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dulamea AO, Sirbu-Boeti MP, Bleotu C, Dragu D, Moldovan L, Lupescu I, Comi G. Autologous mesenchymal stem cells applied on the pressure ulcers had produced a surprising outcome in a severe case of neuromyelitis optica. Neural Regen Res. 2015 Nov;10(11):1841-5. doi: 10.4103/1673-5374.165325. PMID 26807122
- [Background] Xu H, Jiang W, Li X, Jiang J, Afridi SK, Deng L, Li R, Luo E, Zhang Z, Huang YA, Cui Y, So KF, Chen H, Qiu W, Tang C. hUC-MSCs-derived MFGE8 ameliorates locomotor dysfunction via inhibition of ITGB3/ NF-kappaB signaling in an NMO mouse model. NPJ Regen Med. 2024 Jan 20;9(1):4. doi: 10.1038/s41536-024-00349-z. PMID 38242900